CLINICAL TRIAL: NCT06685328
Title: Clinical Study of Minimal Posterior Pole Vitrectomy and Fixing the Inverted Inner Limiting Membrane Flap with Sodium Hyaluronate Gel for Macular Hole
Brief Title: Minimal Vitrectomy and ILM Flap with Sodium Hyaluronate Gel for MH
Acronym: ILM MH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jie Zhong (Other)
Responsible Party: Sponsor-Investigator, Jie Zhong, chief physician, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-598
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Macular Hole; Macular Hole Surgery; Idiopathic Macular Hole; Macular Hole of Left Eye (Disorder); Macular Hole of Right Eye (Disorder)
Keywords: macular hole; inner limiting membrane flap; sodium hyaluronate gel; minimal posterior pole vitrectomy
MeSH Terms: conditions — Retinal Perforations | interventions — Surgical Flaps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- minimal posterior pole vitrectomy (Experimental): Patients undergo minimal posterior pole vitrectomy with tearing of the internal limiting membrane and its folding to cover the macular hole, injection of perfluorocarbon liquid to isolate the balanced salt solution, injection of sodium hyaluronate gel under the perfluorocarbon liquid to cover the folded internal limiting membrane, replacement of the perfluorocarbon liquid and filling of the vitreous cavity with the balanced salt solution and postoperative supine position for 24 hours.
  Interventions: Procedure: minimal posterior pole vitrectomy combined with a sodium hyaluronate gel-covered internal limiting membrane(ILM) flap with balanced saline filling and postoperative supine position
- conventional vitrectomy (Other): Patient undergo conventional vitrectomy with tearing of the inner limiting membrane and flipping to cover the macular hole, gas-liquid exchange and sterile air to fill the vitreous cavity, keeping standard prone position for three days postoperatively.
  Interventions: Procedure: Conventional vitrectomy combined with inner limiting membrane flap flip coverage with sterile air filling and postoperative prone position

INTERVENTIONS:
Procedure: minimal posterior pole vitrectomy combined with a sodium hyaluronate gel-covered internal limiting membrane(ILM) flap with balanced saline filling and postoperative supine position — Vitrectomy of the posterior pole within the vascular arch was performed by a standard 25G ciliary flattening three-way tract procedure, followed by injection of a small amount of tretinoin suspension (TA) to mark the posterior vitreous cortex, which was excised. The inner limiting membrane (ILM) of the macular surface was stained with indocyanine green (ICG, 2.5 mg/ml), and the ILM around the hole was peeled off, leaving a semicircular piece of ILM attached to the hole, and then the single ILM flap was folded and covered with MH. 0.2 to 0.3 mL of hyaluronic acid gel (Bausch & Lomb, Iviz) was injected over the inverted ILM flap using perfluorocarbon liquid for complete coverage. The perfluorocarbon liquid was aspirated. Postoperatively, the patient was advised to remain in a non-emergent supine position for 24 hours.
  Arms: minimal posterior pole vitrectomy
Procedure: Conventional vitrectomy combined with inner limiting membrane flap flip coverage with sterile air filling and postoperative prone position — A standard 25G ciliary flattening three-way tract procedure was taken to perform posterior and midperipheral vitrectomy, followed by injection of a small amount of tretinoin (TA) to label the posterior vitreous cortex and excision of the posterior vitreous cortex within the vascular arch. The ILM on the macular surface was stained with indocyanine green (ICG, 2.5 mg/ml), and the peripapillary ILM was peeled off with forceps, leaving a semicircular piece of ILM attached to the foramen ovale, and the individual ILM flaps were then turned over and covered with MH. Air-liquid exchange was then performed and subsequent surgery was routinely performed according to existing surgical concepts. Ultrasonic emulsification and IOL implantation were selectively performed depending on the extent of the cataract and the patient's surgical needs. Antibiotic ointment is applied at the end of the procedure. After surgery, patients were advised to remain in strict prone position for 3 days.
  Arms: conventional vitrectomy

SUMMARY:
The purpose of this clinical trial is to compare the prognostic validity of two different surgical approaches: minimal posterior pole vitrectomy combined with a sodium hyaluronate gel-covered internal limiting membrane(ILM) flap with balanced saline filling and postoperative supine position, versus conventional vitrectomy combined with ILM flap flap coverage with sterile air filling and postoperative prone position.

The main question it aims to answer is:

Whether patients with macular hole have the same or even better prognosis with minimal posterior pole vitrectomy combined with sodium hyaluronate gel covered flip ILM flap accompanied by balanced salt solution filling accompanied by postoperative supine position than with conventional macular hole surgery.

Participants will:

The control group undergoes conventional vitrectomy combined with internal limbal flap coverage accompanied by sterile air filling of the vitreous cavity and three days of postoperative surgery in strict supine position. The study group undergoes minimal posterior pole vitrectomy combined with sodium hyaluronate gel-assisted flap of the inner border membrane accompanied by 24 hours of postoperative surgical treatment in a non-strict supine position.

Participants of this study come to Sichuan Provincial People's Hospital for follow-up examinations at 1 day, 3 days, 1 week, 1 month, 3 months, and 6 months postoperatively in the 23rd clinic of the Sichuan Provincial People's Hospital for review of visual acuity, intraocular pressure, fundus photography, optical coherence tomography angiography, microfluidic field of view (at 6 months postoperatively), and slit-lamp examination.

DETAILED DESCRIPTION:
Macular hole is a tissue defect that occurs from the inner limiting membrane of the retina to the photoreceptor layer in the macula, severely compromising the patient's central vision. Currently, the standard of care for macular holes is complete vitrectomy combined with stripping, plugging, or flipping of the inner limiting membrane to cover the macular hole, followed by tamponade with prolonged gas or filtered air. After surgery, patients are usually required to remain in a supine position for days to weeks, which is extremely stressful. Despite the effectiveness of current methods, there is still room for thought and improvement.

Given the potential drawbacks of the current mainstream surgery, one investigator developed a minimal posterior pole vitrectomy combined with a sodium hyaluronate gel-assisted flip inner border flap technique for macular hole repair that eliminates the need for prolonged gas or filtered air tamponade and the need for patients to remain in the face-down position for long periods postoperatively. Primary healing was achieved in all postoperative macular holes. However, existing studies have small sample sizes and irregular follow-up times.

In this project, the researchers plan to investigate the prognostic effects of this minimal posterior pole vitrectomy combined with sodium hyaluronate gel-assisted flap with non-strict supine postoperative position for 24 hours and traditional vitrectomy combined with flap covering with sterile air-filled vitreous cavity and strict prone postoperative position for three days on the prognosis of macular holes, and to investigate the therapeutic effects of different surgical methods on macular holes and provide a new idea for the surgical treatment of macular holes. To provide new ideas for the surgical treatment of macular hole.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with idiopathic macular hole and 250 μm ≤ aperture size ≤ 800 μm, with clinical diagnosis based on visual acuity testing, fundus photography, and swept optical coherence tomography/optical coherence tomography angiography (SS-OCT/OCTA)
* Age ≥18 years, gender not restricted
* 22 mm ≤ eye axis ≤ 26 mm
* Patients who can cooperate with accurate microperimetry testing
* Individuals who are able to follow up at the time specified by the researcher

Exclusion Criteria:

* Coexisting active eyelid or appendage infections
* Coexisting ocular pathology other than cataract that affects vision (e.g., retinal detachment or proliferative vitreoretinopathy; diabetic retinopathy; retinal vascular occlusion; uveitis; ocular tumors; glaucoma)
* patients who refused to be randomized
* Other relevant medical history such as cranial brain disease, systemic immune system disease, etc.
* Those who have received medical or surgical treatment other than myopia and cataract in the study eye within the previous 12 months
* Other patients who, in the opinion of the investigator, should be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
postoperative best corrected visual acuity | 1 day, 3 days, 1 week, 1 month, 3 months, 6 months after surgery
  Testing patients' visual function through the visual acuity chart

SECONDARY OUTCOMES:
The time point at which best corrected visual acuity is achieved | 1 day, 3 days, 1 week, 1 month, 3 months, 6 months after surgery
Anatomic closure rate at 6 months postoperatively | 1 day, 3 days, 1 week, 1 month, 3 months, 6 months after surgery
  Evaluate the anatomical structure of the macular area through OCT/OCTA. Recording the proportion of achieving type 1 closure(1A: reconstruction of all retinal layers; 1B outer layer disruption; 1C inner layer disruption) and time point of achieving type 1 closure
Postoperative cataract progression rates in two surgical modalities | 1 day, 3 days, 1 week, 1 month, 3 months, 6 months after surgery
  If the patient have no or mild preoperative cataract, the researchers will observe the rate of postoperative cataract progression in both groups; if the patient have moderate to severe cataract, the researchers will perform cataract surgery at the same time as the macular hole surgery.
Proportion of postoperative displacement of the internal limiting membrane in the two surgical modalities | 1 day, 3 days, 1 week, 1 month, 3 months, 6 months after surgery
  Evaluate the anatomical structure of the macular area through OCT/OCTA
Microperimetry changes: microperimetry at 6 months postoperatively | 6 months after surgery
  Assess macular sensitivity via microperimetry
Incidence of adverse events | Within 6 months after surgery
  e.g., high intraocular pressure, retinal detachment, hemorrhage, cataract worsening, and infection

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes